CLINICAL TRIAL: NCT00355784
Title: Growth Hormone as a Determinant of Weight Regulation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, JEFFREY F HOROWITZ, Associate Professor, Movement Science, School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R01DK071955-01 (NIH); R01DK071955 (NIH)
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Results first posted 2013-07-22 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Obesity
Keywords: growth hormone; overfeeding; energy expenditure; protein metabolism; lipid metabolism
MeSH Terms: conditions — Obesity

ARMS (3):
- Control (Other): 9 non-obese (initial body mass index 23.5 +/- 0.3 kg/m2), weight stable, relatively sedentary (physical activity </- 2h/week), healthy adults not taking any medications were admitted to the hospital for 2 weeks during which time they ate ~4000 kcal/day and their plasma growth hormone concentration was allowed to decline naturally.
  Interventions: Other: overfeeding
- Growth Hormone Treatment (Experimental): 8 non-obese (initial body mass index 23.5 +/- 0.3 kg/m2), weight stable, relatively sedentary (physical activity </- 2h/week), healthy adults not taking any medications were admitted to the hospital for 2 weeks during which time they ate ~4000 kcal/day and received exogenous growth hormone treatment administered in 4 daily injections to mimic physiological growth hormone secretion throughout the 2-week overeating period.
  Interventions: Other: overfeeding; Drug: growth hormone treatment
- High Growth Hormone Treatment (Experimental): 5 non-obese (initial body mass index 23.5 +/- 0.3 kg/m2), weight stable, relatively sedentary (physical activity </- 2h/week), healthy adults not taking any medications were admitted to the hospital for 2 weeks during which time they ate ~4000 kcal/day and received a relatively high daily dose of growth hormone.
  Interventions: Other: overfeeding; Drug: growth hormone treatment

INTERVENTIONS:
Other: overfeeding — overfeeding 2000kcals/day above energy requirements for 14d
Drug: growth hormone treatment — growth hormone administrated for 2 weeks (dose = 1.0 mg/m2/d)
  Arms: Growth Hormone Treatment; High Growth Hormone Treatment

SUMMARY:
With the alarming increase in the prevalence of obesity, identifying factors that predispose individuals to weight-gain is of critical importance. Even when caloric intake and physical activity levels are well controlled, susceptibility for weight-gain is heterogeneous. Basal metabolic rate (BMR) represents the largest portion of daily energy expenditure in normal adults, and as such, variability in BMR among individuals can be a major factor in determining the susceptibility for gaining weight. However, factors responsible for this variability in BMR and resistance to weight-gain remain unclear. Our preliminary data indicate that high-normal growth hormone (GH) concentration is associated with resistance to weight-gain in rats when overfed and greater weight-loss in humans when underfed. In addition, the investigators have found that the pulsatility of GH secretion has profound effects on several metabolic processes. Therefore, together these findings suggest that endogenous GH secretion is associated with body weight regulation, and the pulsatility (peak amplitude) of GH secretion, rather than the absolute GH concentration, per se, may be responsible for this effect. Because GH influences many of the key metabolic processes that contribute to BMR (e.g.; protein synthesis, proteolysis, substrate cycling), the investigators anticipate that the resistance to weight-gain in persons with elevated GH concentrations will be associated with an increase in BMR due to acceleration of some or all of these processes. Our overall hypothesis is that increased GH secretion can protect against weight-gain due to an augmentation of major metabolic processes that contribute to BMR. Identifying factors responsible for predisposing individuals to weight-gain will lead to establishing improved methods for reducing the prevalence of obesity.

DETAILED DESCRIPTION:
The susceptibility to gain weight is highly variable even when caloric intake and physical activity are well controlled. Because basal metabolic rate (BMR) represents ~70% of total daily energy expenditure (TDEE), even a small difference in BMR can affect daily energy balance, thereby increasing the susceptibility for gaining weight. Our preliminary data indicate that high-normal growth hormone (GH) secretion is associated with resistance to weight-gain in rats when overfed and greater weight-loss in humans when underfed. Given that GH influences many of the key metabolic processes that contribute to BMR, the investigators hypothesize that persons with high-normal GH will be resistant to weight-gain because of a high BMR, resulting from accelerated rates of these processes. The investigators will measure basal 24h GH secretion and BMR in 106 non-obese men and women. The investigators will also measure protein synthesis, proteolysis, triglyceride/fatty acid cycling (all measured using stable isotope tracer methods) to determine the relationships among these processes, BMR, and GH [Specific Aim 1]. Subjects identified as having "low-normal" (<1.5 ug/L) and "high-normal" (>3 ug/L) 24h GH will then be admitted to the hospital for a 2 wk overfeeding protocol (~2000 kcal/d >TDEE - with restricted physical activity), immediately followed by a 4 wk caloric restriction protocol (~750 kcal/d <TDEE) to compare changes in weight, body composition and intra-abdominal adiposity between these groups that differ markedly in their GH secretion (GH measured before the diet) [Specific Aim 2]. A subset of subjects with low-normal GH will receive intravenous GH throughout the 2 wk overfeeding period at either: 1. a constant rate or 2. as a pulsatile infusion (to mimic endogenous secretion). BMR will be assessed daily and protein synthesis, proteolysis, and triglyceride/fatty acid cycling will be measured at the end of the 2 wks [Specific Aim 3]. The investigators anticipate that a higher GH pulsatility (peak amplitude), rather than elevated GH concentration, per se, will increase protein synthesis, proteolysis, and triglyceride/fatty acid cycling with a resultant increase in BMR and resistance to weight-gain. Identifying factors responsible for predisposing individuals to weight-gain will help combat the alarming rise in the prevalence of obesity.

ELIGIBILITY:
Inclusion Criteria:

Age = 21-35 years Weight stable (< ± 5 pound over past 6 months) Premenopausal (women only) Body mass index 18 - 26 kg/m2 Must be willing to be randomized to receive GH infusion during 2 week Michigan Clinical Research Unit (MCRU) visit

Exclusion Criteria:

* Evidence of metabolic or cardiovascular disease Pregnancy (women only) Hyperlipidemia (fasting plasma triglyceride concentration > 150 mg/dl) Hematocrit < 34% Liver Function test abnormalities participating in a regular exercise program (> 2 h/week) taking any prescription medication (except birth control)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-09; Primary Completion 2011-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F. Horowitz, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were admitted to the Michigan Clinical Research Unit at the University of Michigan Hospital. Subjects were recruited from February 2006-February 2011.
Pre-assignment Details: Before the overeating intervention all subjects were admitted to the hospital for a 2-day experiment to assess their plasma growth hormone and insulin profiles.
Groups:
- High Growth Hormone Treatment: 5 non-obese (initial body mass index 23.5 +/- 0.3 kg/m2), weight stable, relatively sedentary (physical activity </- 2h/week), healthy adults not taking any medications were admitted to the hospital for 2 weeks during which time they ate ~4000 kcal/day and received a relatively high daily dose of growth hormone throughout the 2-week overeating period.
Period: Overall Study
Arm/Group | Control | Growth Hormone Treatment | High Growth Hormone Treatment
Started | 9 | 8 | 7
Completed | 9 | 8 | 5
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Growth Hormone Treatment | High Growth Hormone Treatment | Total
Number analyzed (Participants) | 9 | 8 | 5 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 5 | 22
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (1.2) | 23.1 (1.0) | 24.9 (1.9) | 24.4 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 7 | 7 | 4 | 18
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Average Plasma Growth Hormone Concentration
Time Frame: 2 weeks
Population: per protocol
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Control (CON): 9 non-obese (initial body mass index 23.5 +/- 0.3 kg/m2), weight stable, relatively sedentary (physical activity </- 2h/week), healthy adults not taking any medications were admitted to the hospital for 2 weeks during which time they ate ~4000 kcal/day and their plasma growth hormone concentration was allowed to decline naturally.
- Growth Hormone Treatment (GHT): 8 non-obese (initial body mass index 23.5 +/- 0.3 kg/m2), weight stable, relatively sedentary (physical activity </- 2h/week), healthy adults not taking any medications were admitted to the hospital for 2 weeks during which time they ate ~4000 kcal/day and received exogenous growth hormone treatment administered in 4 daily injections to mimic physiological growth hormone secretion throughout the 2-week overeating period.
- High Growth Hormone Treatment (High-GHT): 5 non-obese (initial body mass index 23.5 +/- 0.3 kg/m2), weight stable, relatively sedentary (physical activity </- 2h/week), healthy adults not taking any medications were admitted to the hospital for 2 weeks during which time they ate ~4000 kcal/day and received a relatively high daily dose of growth hormone throughout the 2-week overeating period.
Arm/Group | Control (CON) | Growth Hormone Treatment (GHT) | High Growth Hormone Treatment (High-GHT)
Number analyzed (Participants) | 9 | 8 | 5
ng/mL | 0.4 (0.1) | 1.2 (0.1) | 4.1 (0.3)

2. Primary Outcome: Changes in Body Weight
Time Frame: 2 weeks
Population: per protocol
Measure: Mean (Standard Error); unit: kg
Arm/Group | Control (CON) | Growth Hormone Treatment (GHT) | High Growth Hormone Treatment (High-GHT)
Number analyzed (Participants) | 9 | 8 | 5
kg | 2.4 (0.6) | 3.6 (0.6) | 3.1 (0.7)

3. Primary Outcome: Baseline Whole Body Protein Turnover
Description: Whole body proteolytic rate (Leucine Ra)
Time Frame: baseline
Population: per protocol
Measure: Mean (Standard Error); unit: μmol/kg fat free mass/min)
Arm/Group | Control (CON) | Growth Hormone Treatment (GHT) | High Growth Hormone Treatment (High-GHT)
Number analyzed (Participants) | 9 | 8 | 5
μmol/kg fat free mass/min) | 2.1 (0.1) | 1.9 (0.1) | 1.6 (0.1)

4. Primary Outcome: Baseline Skeletal Muscle Protein Synthesis
Description: after an overnight fast
Time Frame: baseline
Population: per protocol
Measure: Mean (Standard Error); unit: skeletal muscle protein%/hour
Arm/Group | Control (CON) | Growth Hormone Treatment (GHT) | High Growth Hormone Treatment (High-GHT)
Number analyzed (Participants) | 9 | 8 | 5
skeletal muscle protein%/hour | 0.043 (0.009) | 0.047 (0.011) | 0.033 (0.006)

5. Primary Outcome: Lipolytic Rate
Time Frame: 2 weeks
Population: per protocol
Measure: Mean (Standard Error); unit: µmol/min
Arm/Group | Control (CON) | Growth Hormone Treatment (GHT) | High Growth Hormone Treatment (High-GHT)
Number analyzed (Participants) | 9 | 8 | 5
µmol/min | 180 (19) | 200 (20) | 195 (25)

6. Primary Outcome: Whole Body Protein Turnover After 2 Week Intervention
Description: whole body proteolytic rate (leucine Ra)
Time Frame: 2 weeks
Population: per protocol
Measure: Mean (Standard Error); unit: µmol/kg fat free mass/min
Arm/Group | Control (CON) | Growth Hormone Treatment (GHT) | High Growth Hormone Treatment (High-GHT)
Number analyzed (Participants) | 9 | 8 | 5
µmol/kg fat free mass/min | 2.8 (0.2) | 2.3 (0.1) | 1.9 (0.1)

7. Primary Outcome: 2 Week Skeletal Muscle Protein Synthesis
Description: after an overnight fast
Time Frame: 2 weeks
Population: per protocol
Measure: Mean (Standard Error); unit: skeletal muscle protein%/hour
Arm/Group | Control (CON) | Growth Hormone Treatment (GHT) | High Growth Hormone Treatment (High-GHT)
Number analyzed (Participants) | 9 | 8 | 5
skeletal muscle protein%/hour | 0.063 (0.015) | 0.062 (0.018) | 0.082 (0.011)

8. Primary Outcome: Changes in Fat Mass
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: kg
Arm/Group | Control (CON) | Growth Hormone Treatment (GHT) | High Growth Hormone Treatment (High-GHT)
Number analyzed (Participants) | 9 | 8 | 5
kg | 1.6 (0.3) | 1.7 (0.2) | 1.1 (0.3)

9. Primary Outcome: Changes in Fat-free Mass
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: kg
Arm/Group | Control (CON) | Growth Hormone Treatment (GHT) | High Growth Hormone Treatment (High-GHT)
Number analyzed (Participants) | 9 | 8 | 5
kg | 0.7 (0.3) | 2.2 (0.3) | 2.3 (0.6)

ADVERSE EVENTS:
Arm/Group | Control (CON) | Growth Hormone Treatment (GHT) | High Growth Hormone Treatment (High-GHT)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 1/9 | 0/8 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (CON) (N=9) | Growth Hormone Treatment (GHT) (N=8) | High Growth Hormone Treatment (High-GHT) (N=5)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Control subject was admitted on 5/7/07. At noon on 5/15, the subject requested to withdraw from the study due to dislike of the food and nausea. Upon follow-up the subject reported that the nausea had resolved.

LIMITATIONS AND CAVEATS:
The short duration of our intervention was a limitation. The metabolic measurements that were performed in the postabsorptive state was a limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes